CLINICAL TRIAL: NCT06349434
Title: The Utilization Effects of Powered Wearable Orthotics in Improving Upper Extremity Function and ADL in Persons With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Ghaith J. Androwis, Ph.D., Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R-1215-23
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: SCI - Spinal Cord Injury; Upper Extremity Dysfunction; Upper Extremity Problem
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MyoPro (Experimental): Receiving MyoMo training in-clinic for 6 weeks, and continuing MyoMo training in-clinic and at home for another 6 weeks.
  Interventions: Device: MyoMo
- Control (Active Comparator): Receiving conventional therapy in-clinic and using their prescribed static brace (or others) for 6 weeks, and continuing the conventional therapy in-clinic and home using their prescribed static brace (or others) at home for 6 weeks.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Device: MyoMo — To evaluate the usefulness of extended utilization of an upper extremity assistive device, called (MyoPro) in improving upper extremity (UE) activities in people with spinal cord injury (SCI).
  Arms: MyoPro
Other: conventional therapy — To evaluate the usefulness of extended conventional therapy compared to the utilization of an upper extremity assistive device called (MyoPro) in improving upper extremity (UE) activities in people with spinal cord injury.
  Arms: Control

SUMMARY:
To evaluate the usefulness of an upper extremity assistive device, called (MyoPro) in improving upper extremity activities in people with incomplete spinal cord injury. The Department of Defense is supporting this study.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a medically complex and life-disrupting condition. Each year in the United States, it is estimated that 17,700 new traumatic SCI cases are reported, including many active service men and women, and veterans. About half of those, the injury involve some part of the arm and hand, representing significant disability and dependence for those patients and their families. When arms/hands are impaired, the patient's quality of life and level of independence are reduced. The proposed RCT investigation will evaluate the long-term effects of the UE-MPWO (MyoPro) in ameliorating wrist/hand/UE movement capability, and increasing ADL and quality of life in people with SCI. This MyoPro orthosis can assist elbow and hand function with built-in motors that are activated by patients' intended motion, as represented by the residue voluntary muscle activities detected by the device's sensors.

The impact of the data generated from this clinical trial investigation should advance the application of new orthotic and prosthetic technologies to treating disabilities as a result of injuries or diseases such as SCI and promote home and community uses of the technologies to improve daily function and independence. The study would also advance scientific knowledge regarding neural changes occurring in the nervous system by application of the technology. The learned knowledge from this investigation will further justify the utilization of such an orthotic technology for individuals with SCI.

Beyond the common therapeutic benefits of upper extremity motor function rehabilitation and assistance for daily living provided with utilization of the MyoPro orthotic device, there may be additional benefits including improvements in quality of life and activity of daily living due to recovered function by using the device. The clinical trial investigation described in this application would provide clinicians and therapists with an initial, but stronger basis for integrating such an orthosis into regimens for managing upper extremity impairments in persons with SCI. This would represent a significant improvement to the existing paradigms of treating hand/arm disabilities in persons with SCI. The benefits, for the patients and society (including the VA community), of utilizing such an orthotic device during daily activities at home and in the community far outweigh the minimal risks associated with this FDA-approved orthosis, particularly as those minimal risks have been minimized by using sound research methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Be between ages 18-80
* Be able to activate certain muscles in my arm and forearm on my own a sufficient amount as measured by EMG amplitude. This will be determined by the study OT/PT.
* Be diagnosed with spinal cord injury (SCI) with level C1-C8 and ASIA Impairment Scale (AIS) C or D, as determined by study staff. If I have not had an exam to determine my injury level and impairment scale recently, I may participate in an examination of my sensation and strength in my arms, legs, trunk and rectum as was done in the hospital soon after my injury.
* Be at least 1-year post injury
* Have sufficient ability to move my shoulder (active shoulder flexion of 30 degrees and active shoulder abduction 20 degrees), as determined by study staff
* Be medically stable
* Have sufficient learning and memory abilities and abilities to communicate in English to be able to participate and follow directions during my rehabilitation
* Continue to take all prescribed medication (e.g., oral or via pump baclofen) without any dosing changes
* Be able to tolerate functional tasks for 60 minutes with periodic rests without excessive fatigue
* Have minimal strength in the muscles that bend and straighten my elbow, as determined by study staff
* Have full range of motion in my elbow when it is moved by the study therapist

Exclusion Criteria:

* Be younger than 18 years old or older than 80
* Have excessive pain in my arm, wrist, or hand that limits providing rehabilitation
* Have excessive spasticity in my elbow or wrist, as determined by study staff
* Be participating in any experimental rehabilitation or drug studies
* Have history of nervous system disorder other than SCI
* Have difficulty following multiple step directions
* Have severe cognitive or psychiatric problems might be contraindications to start training.
* Have skin issues or severe sensory deficits that would prevent wearing the Myo-Pro device safely
* Be pregnant
* Have other conditions or circumstances that, in the opinion of the investigators, would affect the safety or effectiveness of the training in which I would participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
GRASSP | Approximately 36 weeks
  Assessment of the Hand in Tetraplegia Using the Graded Redefined Assessment of Strength Sensibility and Prehension Upper Extremity (UE) Function in Persons with Tetraplegia Relationships Between Strength, Capacity and the Spinal Cord Independence Measure.
  Total score's minimum and maximum values are between 0 to 116 and higher scores indicate better/improved outcomes.
Range of motion of hands and arms | Approximately 36 weeks
  Movement of upper extremity is measured using small sensors that are able to record joints' angles. These sensors are placed on participant's skin via double sticky tape.
  Participants will be asked to move their hand and forearm while the elbow, wrist and hand joint angles are measured.
Muscle strength measurement | Approximately 36 weeks
  during movements of upper extremities muscle strength is measured using small and light weight surface electromyography sensors which are placed on the participant's skin via double stick tape.
  Participants will be asked to move their hand and forearm while the muscle strength is measured.

SECONDARY OUTCOMES:
Spasticity measurement | Approximately 36 weeks
  Spasticity measurements of upper and lower extremities using the Modified Ashworth scale (MAS).
  The MAS scores range between 0 to 4. A higher score signifies larger level of spasticity and a lower score indicates smaller level of spasticity. scores are as follows:
  0: No increase in muscle tone
  Slight increase in muscle tone 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion More marked increase in muscle tone through most of the range of motion. Considerable increase in muscle tone, passive movement difficult Affected part(s) rigid in flexion or extension
Brain signals measurement | Approximately 36 weeks
  Measurements of brain signals is done using a cap and electrodes that would be placed on the participant's head using surface electrodes.
  Participants will be asked to move their extremities while brain signals are measured.
CUE-Q | Approximately 36 weeks
  The Capabilities of Upper Extremity Test (a list of questionnaire based evaluation).
  Scores range between 0 to 4, and higher scores indicates better ability outcome for reaching or lifting the upper limb.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided